CLINICAL TRIAL: NCT01477710
Title: Ability of Caregivers to Provide Ventilation With the SAVe Resuscitator in a Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rich Branson, M.D., Professor Emeritus, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Branson-2010-01
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pre-hospital Ventilation
Keywords: Mechanical ventilation; Tidal volume; Respiratory rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hold Mask (Active Comparator): The clinician will connect a SAVe ventilator to a face mask and hold the mask in place on the mannequin with two hands while maintaining the airway on the correct position for 10 minutes.
  Interventions: Procedure: Hold mask
- Strap Mask (Active Comparator): The clinician will attach the face mask to the mannequin using the mask and mask strap included in the ventilator kit for 10 minutes
  Interventions: Procedure: Strap Mask
- Airway (Active Comparator): The clinician will blindly insert a supralaryngeal airway (the King lT) and connect the SAVe ventilator to the connector and provide ventilation for 10 minutes.
  Interventions: Procedure: Airway

INTERVENTIONS:
Procedure: Hold mask — The clinician will connect a SAVe ventilator to a face mask and hold the mask in place on the mannequin with two hands while maintaining the airway on the correct position for 10 minutes.
  Arms: Hold Mask
Procedure: Strap Mask — The clinician will attach the face mask to the mannequin using the mask and mask strap included in the ventilator kit for 10 minutes
  Arms: Strap Mask
Procedure: Airway — The clinician will blindly insert a supralaryngeal airway (the King lT) and connect the SAVe ventilator to the connector and provide ventilation for 10 minutes.
  Arms: Airway

SUMMARY:
This study will compare three methods of delivering mechanical ventilation using a test lung. Ventilation will be delivered using (1) a mask held in place by a caregiver, (2) a mask strapped to the model using a securing device, and (3) a supraglottic airway. Endpoints include respiratory rate and tidal volume.

DETAILED DESCRIPTION:
To evaluate the ability of caregivers to provide adequate ventilation (respiratory rate and tidal volume) in a model of the upper airway and lungs. Ventilation will be delivered while the mask is held in place by the caregiver, with the mask strapped to the model using the securing device provided with the ventilator, and following placement of a supraglottic airway.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Nurse, respiratory therapist, or physician
* involved in the care of patients requiring ventilation and airway management

Exclusion Criteria:

-

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Branson, MSc RRT, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects (registered nurses, respiratory therapists, and physicians) volunteered to participate and signed informed consent documents.
Groups:
- All Participants: Each participant will perform 3 tasks -- in the same order. First, the clinician will connect a SAVe ventilator to a face mask and hold the mask in place on the mannequin with two hands while maintaining the airway on the correct position for 10 minutes. Next, the clinician will attach the face mask to the mannequin using the mask and mask strap included in the ventilator kit for 10 minutes. Finally, the clinician will blindly insert a supralaryngeal airway (the King lT) and connect the SAVe ventilator to the connector and provide ventilation for 10 minutes.
Period: Overall Study
Arm/Group | All Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each clinician will connect a SAVe ventilator to a face mask and hold the mask in place on the mannequin with two hands while maintaining the airway on the correct position for 10 minutes. Then, each will attach the face mask to the mannequin using the mask and mask strap included in the ventilator kit for 10 minutes. Finally, each will blindly insert a supralaryngeal airway (the King lT) and connect the SAVe ventilator to the connector and provide ventilation for 10 minutes.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Tidal Volume
Description: Nurses, respiratory therapists, and physicians will provide mechanical ventilation to a test instrument using three techniques of airway management. Each participant will ventilate the model using each technique for 10 minutes, in random order. During each period, the breath-to-breath tidal volume, respiratory rate, inspiratory flow, inspiratory time, and airway pressure will be recorded.
Time Frame: 10 minutes per technique, for a total of 30 minutes per participant
Measure: Mean (Standard Error); unit: milliliters (mL)
Groups:
- Hold Mask: Mask is held in place by caregiver.
- Strap Mask: Mask is strapped to model using a securing device
- Airway: Using a supraglottic airway
Arm/Group | Hold Mask | Strap Mask | Airway
Number analyzed (Participants) | 30 | 30 | 30
milliliters (mL) | 341.8 (17.7) | 27.5 (17.7) | 604.1 (17.7)
Statistical Analysis 1: Comparison: Hold Mask vs Strap Mask vs Airway; Using ANOVA, pairwise comparisons of treatment means were made using a Tukey adjustment for multiple comparisons; Test type: Superiority or Other; p < 0.0001, ANOVA — This p-value is for the omnibus F-test of between-treatment differences in tidal volume; The p-value for the omnibus F-test was <0.0001; ANOVA F-value = 266.39
Statistical Analysis 2: Comparison: Hold Mask vs Strap Mask; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 314.4, 95% CI [264.7 to 364.1]
Statistical Analysis 3: Comparison: Strap Mask vs Airway; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 576.6, 95% CI 2-sided [526.9 to 626.3], Standard Error of Mean 25.0
Statistical Analysis 4: Comparison: Hold Mask vs Airway; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 262.2, 95% CI 2-sided [212.5 to 312.0], Standard Deviation 25.0

ADVERSE EVENTS:
Arm/Group | Hold Mask | Strap Mask | Airway
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes